All About Me: An Intervention to Ease the Transition to Long-term Care, Build Community, and Improve Quality of Care for Persons with Dementia NCT05516134

Statistical Analysis Plan 7/27/22

The All About Me app will be considered successful if persons with dementia exhibit higher levels of positive engagement/affect and lower levels of negative engagement--as measured by the Menorah Park Engagement Scale (MPES))--during the intervention, as compared to standard programming at baseline. First, multiple observations of participants will be taken at both baseline and treatment on both scales. Then, means will be calculated for each participant for each item (on the MPES). Then, we will conduct a paired sample *t*-test to determine whether there are significant differences from baseline to treatment. We will also conduct paired sample *t*-tests to examine whether participants exhibit an improvement in the Dementia-Related Quality of Life Scale (DEMQOL), Geriatric Depression Scale – Short Form (GDS-SF), and Neuropsychiatric Inventory – Nursing Home (NPI-NH).